CLINICAL TRIAL: NCT02646319
Title: A Pilot Study of a Rapid Access Platform for Investigational Drugs (RAPID) in Advanced Cancers
Brief Title: Nanoparticle Albumin-Bound Rapamycin in Treating Patients With Advanced Cancer With mTOR Mutations
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1313; NCI-2015-02151 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1313 (Other: Mayo Clinic in Arizona); P30CA015083 (NIH)
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2018-06

CONDITIONS: Advanced Malignant Neoplasm; Cervical Squamous Cell Carcinoma; Endometrial Carcinoma; Malignant Uterine Neoplasm; Recurrent Bladder Carcinoma; Recurrent Breast Carcinoma; Recurrent Cervical Carcinoma; Recurrent Head and Neck Carcinoma; Recurrent Malignant Neoplasm; Recurrent Ovarian Carcinoma; Recurrent Prostate Carcinoma; Recurrent Renal Cell Carcinoma; Solid Neoplasm; Stage III Bladder Cancer; Stage III Prostate Cancer; Stage III Renal Cell Cancer; Stage IIIA Breast Cancer; Stage IIIA Cervical Cancer; Stage IIIA Ovarian Cancer; Stage IIIB Breast Cancer; Stage IIIB Cervical Cancer; Stage IIIB Ovarian Cancer; Stage IIIC Breast Cancer; Stage IIIC Ovarian Cancer; Stage IV Breast Cancer; Stage IV Ovarian Cancer; Stage IV Prostate Cancer; Stage IV Renal Cell Cancer; Stage IVA Bladder Cancer; Stage IVA Cervical Cancer; Stage IVB Bladder Cancer; Stage IVB Cervical Cancer
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms; Urinary Bladder Neoplasms; Breast Neoplasms; Uterine Cervical Neoplasms; Recurrence; Ovarian Neoplasms; Prostatic Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nanoparticle albumin-bound rapamycin) (Experimental): Patients receive nanoparticle albumin-bound rapamycin IV over 30 minutes on days 1 and 8. Treatment repeats every 21 days for 24 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Nanoparticle Albumin-Bound Rapamycin; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nanoparticle Albumin-Bound Rapamycin — Given IV
  Other Names: ABI-009; Nab-Rapamycin
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot trial studies how well nanoparticle albumin-bound rapamycin works in treating patients with cancer that as has spread to other places in the body and usually cannot be cured or controlled with treatment (advanced cancer) and that has an abnormality in a protein called mechanistic target of rapamycin (mTOR). Patients with this mutation are identified by genetic testing. Patients then receive nanoparticle albumin-bound rapamycin, which may stop the growth of cancer cells by blocking the mTOR enzyme, which is needed for cell growth and multiplication. Using treatments that target a patient's specific mutation may be a more effective treatment than the standard of care treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate efficacy of groups of patients defined by disease type, genomic aberration and treatment regimen.

II. To assess the confirmed response rate of nanoparticle albumin-bound rapamycin (nab-rapamycin) in mTOR aberrant advanced cancers. (Sub-protocol Arm A)

SECONDARY OBJECTIVES:

I. To estimate other clinical outcomes (e.g., progression-free and overall survival) of groups of patients defined by disease type, genomic aberration and treatment regimen.

II. To describe the adverse event profile of each regimen. III. To assess the clinical benefit rate of nab-rapamycin in mTOR aberrant advanced cancers. (Sub-protocol Arm A).

IV. To estimate progression-free survival (specifically at 6 months) and overall survival of these patients. (Sub-protocol Arm A) V. To estimate the adverse event profile of nab-rapamycin. (Sub-protocol Arm A)

TERTIARY OBJECTIVES:

I. To describe patient health-related quality of life (HRQOL) and symptoms using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core (QLQ-C)30 in groups of patients defined by disease type and/or treatment regimen and to correlative HRQOL/symptoms with genomic markers.

II. To assess the rate of individual mTOR pathway aberrations and assess the association between individual mTOR pathway aberrations and clinical outcome both across disease indications and within disease indications. (Sub-protocol Arm A)

OUTLINE:

Patients receive nanoparticle albumin-bound rapamycin intravenously (IV) over 30 minutes on days 1 and 8. Treatment repeats every 21 days for 24 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of cancer which is now not amenable to curative standard treatment options
* Patient must have received at least 1 prior standard therapy for their disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Ability to provide informed written consent
* Willing to return to enrolling institution for follow-up (active monitoring phase of the study); Note: During the active monitoring phase of a study (i.e., active treatment), participants must be willing to return to the consenting institution for follow-up
* Life expectancy >= 84 days (3 months)
* Identification of a drug target/targets through molecular profiling performed as a part of routine clinical care and treatment recommendation by the Mayo Clinic Genomics Tumor Board (GTB); NOTE: If profile matches more than 1 treatment arm, final decision for treatment arm assignment to be made by patients treating physician; it will be required for the genomic aberration to be identified through a test in a Clinical Laboratory Improvement Amendments (CLIA) workflow; assays used will range from single gene abnormalities (e.g. fluorescent in situ hybridization [FISH] for human epidermal growth factor receptor 2 [ERBB2] amplifications) to next generation sequencing based gene panels (Foundation One®) to more comprehensive assays such as whole exome sequencing; the Mayo Clinic GTB will serve as the centralized point of data synthesis to allow for assessment of molecular profiling accomplished through a heterogeneous array of tests
* Date of Mayo Clinic Genomics Tumor Board review =< 3 months prior to registration
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria (for solid tumors) or equivalent criteria (for patients with non-solid tumor malignancies)
* Patient meets all sub-protocol specific criteria of each applicable sub-protocol
* Ability to complete questionnaire(s) by themselves or with assistance
* SUB-PROTOCOL AIM A: Histological confirmation of renal cell carcinoma, head and neck cancer, endometrial cancer, breast cancer, ovarian cancer, prostate cancer, squamous cell cervical or uterine cancer, or bladder cancer
* SUB-PROTOCOL AIM A: Confirmation of advanced cancer with mTOR pathway aberrations as determined through routine clinical care using pathway aberrations performed in a CLIA certified laboratory; cancer genomic profiling tests incorporating next generation sequencing from archival formalin-fixed paraffin-embedded tissue (FFPE) are validated with sensitivities and specificities of 99% and 99%, respectively; in the assay, hybrid-capture-selected deoxyribonucleic acid (DNA) libraries are sequenced to depths targeting > 500 × coverage by non-polymerase chain reaction (PCR) duplicate read pairs, with > 99% of exons at coverage > 100 ×); multiplatform profiling may include immunohistochemistry and in situ hybridization methods with previously established negative/positive cutoffs performed in a CLIA certified lab; at least one pathway aberration must be identified; these must be confirmed in a CLIA certified lab; the potential mTOR aberrations that could be identified are listed below, please note that this list is not all inclusive; if a CLIA validated report lists an mTOR pathway inhibitor as a target drug for a genetic aberration, then it can be considered eligible for the purposes of this study; v-akt murine thymoma viral oncogene homolog 1 (AKT1), MTOR, phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA), tuberous sclerosis (TSC)1, TSC2, retrovirus-associated DNA sequence (Ras) homolog enriched in brain (RHEB), serine/threonine kinase 11 (STK11), neurofibromin (NF)1/2
* SUB-PROTOCOL AIM A: Absolute neutrophil count (ANC) >= 1500/mm^3
* SUB-PROTOCOL AIM A: Platelet count >= 100,000/mm^3
* SUB-PROTOCOL AIM A: Hemoglobin >= 9.0 g/dL
* SUB-PROTOCOL AIM A: Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* SUB-PROTOCOL AIM A: Aspartate transaminase (AST); alanine aminotransferase (ALT) =< 1.5 x ULN; NOTE: if subject has tumor involvement in the liver =< 5 X ULN
* SUB-PROTOCOL AIM A: Serum cholesterol =< 350 mg/dL
* SUB-PROTOCOL AIM A: Serum triglyceride =< 300 mg/dL
* SUB-PROTOCOL AIM A: Serum creatinine =< 1.5 x ULN
* SUB-PROTOCOL AIM A: Previously treated patients who have failed, unable to tolerate, or refused other available active therapies
* SUB-PROTOCOL AIM A: Women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (e.g., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test =< 14 days prior to registration and must use two forms of highly effective contraception (also applicable to their partners who are biologically able to conceive)
* SUB-PROTOCOL AIM A: Adequate coagulation function as defined by either of the following criteria:

  * International normalized ratio (INR) =< 1.5 x ULN
  * For subjects receiving warfarin or low molecular weight heparin (LMWH), the subjects must, in the investigator's opinion, be clinically stable with no evidence of active bleeding while receiving anticoagulant therapy; the INR for these patients may exceed 1.5 x ULN if that is the goal of the anticoagulant therapy

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Failure to fully recover from acute, reversible effects of prior chemotherapy (other anti-neoplastic therapy) and radiation therapy to adverse event severity of =< grade 1
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* SUB-PROTOCOL AIM A: Any of the following:

  * Pregnant women
  * Nursing women
  * Women of child-bearing potential, who are biologically able to conceive, or men who are able to father a child, not employing two forms of highly effective contraception

    * Highly effective contraception (e.g., male condom with spermicide, diaphragm with spermicide, intra-uterine device, and total abstinence) must be used by both sexes during the study and must be continued for 6 months after the end of study treatment; Note: Oral, implantable, or injectable hormone contraceptives are not considered effective for this study
* SUB-PROTOCOL AIM A: Any of the following treatments:

  * Chemotherapy within 4 weeks before treatment with nab-rapamycin
  * Hormonal therapy within 4 weeks before treatment with nab-rapamycin (with the exception of leuprolide, degarelix, or goserelin)
  * Immunotherapy within 4 weeks before treatment with nab-rapamycin
  * Radiotherapy within 4 weeks before treatment with nab-rapamycin
  * Treatment with nitrosoureas, mitomycin, or extensive radiotherapy within 6 weeks before treatment with nab-rapamycin
  * Immunosuppressive agents within 3 weeks before treatment with nab-rapamycin (except corticosteroids used as antiemetics)
  * Use of prior mTOR pathway inhibitor therapy
* SUB-PROTOCOL AIM A: Patients with a history of interstitial lung disease and/or pneumonia
* SUB-PROTOCOL AIM A: Receiving any concomitant antitumor therapy or inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4)
* SUB-PROTOCOL AIM A: History of allergic reactions attributed to compounds of similar chemical or biologic composition including macrolide (e.g. azithromycin, clarithromycin, dirithromycin, and erythromycin) and ketolide antibiotics
* SUB-PROTOCOL AIM A: Major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) =< 4 weeks prior to registration or failure to recover from side effects of such surgery; exceptions: port placements, nephrectomy, tumor biopsies, and minor surgeries
* SUB-PROTOCOL AIM A: Concurrent use of any other approved or investigational anticancer agents which would be considered as a treatment for the primary neoplasm
* SUB-PROTOCOL AIM A: Patients with a history of alcoholism, drug addiction or psychotic disorders
* SUB-PROTOCOL AIM A: Uncontrolled diabetes mellitus as defined by hemoglobin A1C (HbA1c) > 8% despite adequate therapy; unstable coronary artery disease or myocardial infarction during preceding 6 months; or hypertension uncontrolled by medication
* SUB-PROTOCOL AIM A: Patients who required therapeutic doses of anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Proportion of confirmed responses, evaluated using the RECIST v1.1 | Up to 21 days
  The proportion of confirmed responses will be estimated by the number of confirmed responses divided by the total number of evaluable patients. An exact binomial confidence interval for the true confirmed response proportion will be calculated. Analysis will be carried out overall and within disease groups where warranted by sample size.

SECONDARY OUTCOMES:
Clinical benefit rate defined as the proportion of patients with a confirmed response or stable disease (complete response+partial response+stable disease) divided by the total number of evaluable patients | Up to 5 years
  An exact binomial confidence interval for the true confirmed clinical benefit rate will be calculated. Analysis will be carried out overall and within disease groups where warranted by sample size.
Incidence of adverse events, using the National Cancer Institute Common Terminology Criteria for Adverse Events v4.0 | Up to 30 days after last dose of study treatment
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration. Analysis will be carried out overall and within disease groups where warranted by sample size.
Survival time | Time from registration to death due to any cause, assessed up to 5 years
  The distribution of survival time will be estimated using the method of Kaplan-Meier. Analysis will be carried out overall and within disease groups where warranted by sample size.
Time to disease progression | Time from registration to the earliest date of documentation of disease progression, assessed up to 5 years
  The distribution of time to progression will be estimated using the method of Kaplan-Meier. The 6-month progression-free rate will be provided. Analysis will be carried out overall and within disease groups where warranted by sample size.

OTHER OUTCOMES:
Quality of life, measured using the EORTC QLQ-C30 | Up to 24 weeks
  Scale score trajectories over time will be examined using stream plots and mean plots with standard deviation error bars overall and by disease group where warranted by sample size. Changes from baseline at each cycle will be statistically tested using paired t-tests, and standardized response means (mean of the change from baseline scores at a given cycle, divided by the standard deviation of the change scores) will be interpreted (after applying Middel's adjustment) using Cohen's cut-offs.
Rate of individual mTOR pathway aberrations | Up to 5 years
  Will be described, and association with confirmed response will be investigated using a Fisher's exact test. Associations with time to progression and overall survival will be investigated using log-rank tests. Analysis will be carried out overall and within disease groups where warranted by sample size.

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Borad, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota